CLINICAL TRIAL: NCT02820948
Title: Effect of Subcutaneous Sterile Vitamin E Ointment on Incisional Surgical-site Infection Following Elective Laparoscopic Colorectal Cancer Surgery
Brief Title: Effect of Vitamin E Ointment on Incisional SSI in Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, David Alias, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC 16-6
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin E ointment application (Experimental): Before the skin stapling and after the subcutaneous irrigation with normal saline, sterile Vitamin E acetate ointment was applied in the subcutaneous tissue; 2 ml were applied in the suprapubic incision and 0.5 ml in the rest of port sites.
  Interventions: Drug: Vitamin E ointment application
- No Vitamin E ointment application (No Intervention): No vitamin E ointment was performed.

INTERVENTIONS:
Drug: Vitamin E ointment application — Before the skin stapling and after the subcutaneous irrigation with normal saline, sterile Vitamin E acetate ointment was applied in the subcutaneous tissue; 2 ml were applied in the suprapubic incision and 0.5 ml in the rest of port sites.
  Other Names: Subcutaneous sterile Vitamin E acetate ointment application
  Arms: Vitamin E ointment application

SUMMARY:
A prospective, randomized study was performed. The patients were randomized into 2 groups: those patients undergoing subcutaneous vitamin E ointment application (Group 1) and those patients who not (Group 2).

Incisional surgical site infection (SSI), microbiological cultures from the infected surgical wounds, postoperative pain and acute phase reactants were investigated.

DETAILED DESCRIPTION:
A prospective, randomized study was performed. The patients were randomized into 2 groups: those patients undergoing a subcutaneous sterile vitamin E acetate ointment application (Group 1) and those patients who did not receive this vitamin E ointment application (Group 2).

Before the skin stapling and after the subcutaneous irrigation with normal saline, sterile Vitamin E acetate ointment (FilmeOft, Hulka SRL, Rovigo, Italy) was applied in the subcutaneous tissue; 2 ml were applied in the suprapubic incision and 0.5 ml in the rest of port sites.

Incisional SSI, microbiological cultures from the infected surgical wounds, postoperative pain was evaluated 24 hours after surgery by means of a Visual Analogic Scale (VAS), ranging from 0 mm (complete absence of pain) to 100 mm (unbearable pain) and acute phase reactants (white cell count (WBC), fibrinogen and C reactive protein) 48 hours after surgery were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal neoplasms and plans to undergo an elective laparoscopic surgery with curative aims

Exclusion Criteria:

* Open surgical approach or conversion to laparotomy
* Performance of a stoma
* Immunodepression status
* Anastomotic leak

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia, Study Director — Fundacion Jimenez Diaz

IPD SHARING:
Plan to Share IPD: Yes
Publication in scientific journal